CLINICAL TRIAL: NCT06187090
Title: The Supplementation Therapy in Autism and Response to Treatment (START) Study
Brief Title: The Supplementation Therapy in Autism and Response to Treatment Study
Acronym: START
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Udine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-DAME 188/2023
Record Dates: First submitted 2023-12-15; First posted 2024-01-02 (Actual); Last update posted 2024-01-02 (Actual); Status verified 2023-12

CONDITIONS: Autism; Autism Spectrum Disorder; Autism Spectrum Disorder High-Functioning; Asperger Syndrome; Depressive Symptoms; Anxiety State
MeSH Terms: conditions — Autistic Disorder; Autism Spectrum Disorder; Asperger Syndrome; Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: 12-week, open-label, investigator-initiated proof-of-concept study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PEA Arm (Experimental)
  Interventions: Dietary Supplement: Oral Ultramicronized-Palmitoylethanolamide (um-PEA; 600 mg per day) in tablet form

INTERVENTIONS:
Dietary Supplement: Oral Ultramicronized-Palmitoylethanolamide (um-PEA; 600 mg per day) in tablet form — Um-PEA is to be taken orally once a day (600 mg per day) around mealtime during the 12-week initial phase of the study. During the 24-week extension phase of the study, the trial medication is to be taken from once a day up to twice a day (600-1200 mg per day), based on clinical judgment of the improvement obtained so far, around mealtime.

SUMMARY:
In addition to the "core" symptoms of ASD (i.e., impaired communication, impaired reciprocal social interaction and restricted, repetitive and stereotyped patterns of behaviors or interests), it is estimated that up to 70% of autistic people present at least one comorbid psychiatric disorder, leading to a deterioration in quality of life, a greater demand for support and worse prognosis and outcome. Anxiety and depressive symptoms would seem to be more present in individuals with Level 1 ASD, requiring their prioritisation against core symptoms. To date, the first-line treatment for autistic patients with comorbid depressive and/or anxiety symptoms is still debated and it is not always clear whether they may or may not benefit from psychotherapeutic and conventional psychopharmacological approaches. As such, growing evidence strengthens the therapeutic potential of the endocannabinoid (eCB) system modulation and of eCB-like compounds.

The aim of this study is to provide a response to an unmet clinical need in this framework of psychic vulnerability by initiating oral therapy with palmitoylethanolamide (PEA), a nutraceutical/food supplement with proven anti-inflammatory and neuroprotective properties.

Indeed, many conditions of psychological distress are thought to be underpinned by systemic inflammatory and/or neuroinflammatory processes, on which PEA has shown remarkable efficacy, including through modulation of the immune response and the interaction between the endocannabinoid system and the gut-microbiota-brain axis.

The trial we are proposing is a 12-week open-label phase 2 study involving the daily intake of PEA 600 mg, at a dosage of 1 tablet/day.

This study will be conducted at the Unit of Psychiatry of Santa Maria della Misericordia Udine University Hospital.

Through this study, we wish to evaluate: the ability of PEA to alleviate symptoms of psychic distress (i.e., anxiety and/or depression) in Level 1 autistic adults; the safety and tolerability of sustained intake of PEA in Level 1 autistic adults; and the biological basis of PEA functioning.

The study involves taking PEA orally once daily (600 mg daily) at the same time as a meal during the initial 12-week phase. Upon completion of the initial phase, subjects will be offered to enter an extension phase of the trial of an additional 24 weeks to assess treatment stability, with the possibility of titration of PEA to 1200 mg daily based on observed clinical compensation. Each participant will be on PEA treatment for up to 36 weeks.

During the course of the study, periodic clinical re-evaluations will be conducted at our Day-Hospital setting.

The trial will unfold through one screening visit, one baseline visit, and two follow-up visits (FUP, 4 weeks and 12 weeks apart). The patient will be administered standardized interviews by a qualified investigating physician; clinical objective examination, collection of blood and urine samples for standard hematochemical investigations, collection of blood and stool samples for analysis of some biological markers of interest, monitoring of adherence to therapy intake, side effects, and adverse effects will also be performed during the follow-up visits. The nutraceutical PEA will be dispensed by the clinical investigators at each follow-up visit.

DETAILED DESCRIPTION:
1. RATIONALE FOR CURRENT STUDY

   The main purpose of the present study is to address a major unmet clinical need for Level 1 autistic individuals with comorbid anxiety and/or depressive symptoms, with respect to a condition of psychic vulnerability not responding to conventional psychopharmacological approaches. We will thus perform an investigator-initiated proof-of-concept study (Phase-2 Pilot Study), with the purpose to examine:

   (i) Palmitoylethanolamide (PEA) ability to alleviate symptoms of psychic distress (i.e., anxiety and/or depression) in Level 1 autistic individuals; (ii) PEA safety and tolerability; (iii) The biological basis of PEA effect.
2. TRIAL OBJECTIVES

   To evaluate:

   (i) The viability of identifying and consenting Level 1 autistic volunteers into a trial with PEA; (ii) The efficacy of PEA in providing relief to anxiety and/or depressive symptoms in Level 1 autistic individuals; (iii) Whether sustained PEA treatment is well tolerated by Level 1 autistic individuals over a period of at least 12 weeks; (iv) The biological mechanisms underpinning PEA beneficial effects in Level 1 autistic individuals (e.g., modulation of the endocannabinoid (eCB) system, immunological response, metabolic fingerprinting, gut microbiome composition).

   2.1. Objective (i) Feasibility questions

   Over the first 12 months from first patient recruited we will assess whether:

   (i) A minimum of 20 eligible volunteers have consented to be enrolled into the study; (ii) At least 80% of recruited patients have completed the 12-week follow-up; Feasibility endpoints (i) Number of subjects giving consent; (ii) Proportion of participants completing the 12-week follow-up.

   2.2. Objective (ii) Research Questions

   Our primary clinical research question is whether PEA added to treatment as usual (TAU) in Level 1 autistic individuals:

   (i) Improves psychic distress (i.e., anxiety and depressive symptoms) to the extent of impacting on levels of self-sufficiency;

   Our secondary clinical research questions are whether PEA added to TAU in Level 1 autistic individuals:

   (ii) Reduces the intensity of anxiety and/or depressive symptoms, with particular regards to the subdomains of somatisation, anxiety and depression; (iii) Improves interpersonal and neurocognitive functioning. Primary endpoints Assessing the global improvement in symptom intensity and psychological distress associated with autism through the Global Score Index (GSI) of the SCL-90-R.

   Secondary endpoints (i) Impact on levels of personal autonomy as measured through the WHODAS 2.0 total score.

   (ii) Severity of anxiety symptoms as assessed using the Hospital Anxiety and Depression Scale (HADS) and the somatisation, anxiety and depression subscales of the SCL-90-R; (iii) Severity of neurocognitive and interpersonal functioning as assessed using the subdomains 1 'cognitive activities' and 4 'interpersonal relationships' of the WHODAS 2.0.

   All the study endpoints for the 12-week clinical trial will be assessed by comparing follow-up (FUP) visits and baseline. For those participants continuing in the 24-week extension phase, change (FUP visit minus baseline) in symptom intensity and psychological distress associated with autism as measured through the GSI of the SCL-90-R and the impact on levels of personal autonomy measured through the WHODAS 2.0 total score will be compared with the group of those willing to discontinue PEA and continue with TAU.

   2.3. Objective (iii) Safety questions We will evaluate if sustained PEA treatment is well tolerated, with minimal side-effects.

   Safety endpoints Incidence of adverse effects during the study period, as measured using the UKU side-effect rating scale.
3. TRIAL DESIGN We will evaluate the study viability through an internal pilot that will assess the ability of the study to identify, consent, and follow up Level 1 autistic volunteers experiencing anxiety and/or depressive symptoms in the study. We propose a 12-week, open-label, investigator-initiated proof of concept study (Phase-2 Pilot Study) of PEA (600 mg/day) for the treatment of psychic distress (i.e., sub-threshold anxiety and/or depressive symptoms) in Level 1 autistic individuals. We plan to enrol 20 young adults diagnosed with Autism Spectrum Disorder (ASD). Those completing the 12-week initial phase, will be proposed to enter a 24-week extension phase to evaluate the clinical stability of treatment, with the possibility of PEA titration to 1200 mg/day based on clinical improvement obtained so far.
4. PARTICIPANTS 4.1. Selection of participants The proposed single-centre study will involve a university clinical research facility in Italy. Participants will be enrolled into the internal pilot, that will progress to the open-label trial. Volunteers who express an interest in the study and are identified as having Level 1 autistic individuals with comorbid anxiety and/or depressive symptoms by their clinical teams will be approached by study researchers and given a patient information sheet. Those who agree to take part in the study will be invited for a screening visit.

   4.2. Heterogeneity in autism spectrum disorder ASD comprises three subgroups of patients based on the severity of symptoms whose classification is based on impairment of social communication and restricted, repetitive behaviour patterns: (i) Level 1 'Support is needed', (ii) Level 2 "Significant support is needed", (iii) Level 3 "Very significant support is needed very significant support'. As the present study was designed to assess the effect of PEA on mentally fragile conditions with interference in the global functioning of autistic individuals, we will focus on subjects with severity level 1, more affected by depressive and anxious symptoms than autistic subjects with higher levels of impairment, requiring a prioritisation of these manifestations compared to core symptoms. Symptoms of psychological distress in ASD individuals, below the threshold of clinical criteria for the diagnosis of a full-blown psychiatric disorder and not requiring the introduction of conventional psychotropic medications, are nevertheless often deserving of an intervention to support their well-being.
5. INTERVENTION 5.1. Trial Medication Oral Palmitoylethanolamide (PEA; 600 mg per day) in tablet form. PEA will be obtained by a pharmaceutical company operating under good manufacturing practice conditions with appropriate certification. The information presented on the labels for PEA will comply with applicable national and local regulations.

   5.2. Dosing Regimen PEA is to be taken orally once a day (600 mg per day) around mealtime during the 12-week initial phase of the study. During the 24-week extension phase of the study, the trial medication is to be taken from once a day up to twice a day (600-1200 mg per day), based on clinical judgment of the improvement obtained so far, around mealtime. Each participant will undergo PEA treatment for a maximum of 36 weeks. The information presented on the labels for the PEA will comply with applicable national and local regulations.

   5.3. Medication Risks Being a food supplement/nutraceutical, PEA can be purchased at pharmacies without a medical prescription. While unknown risks cannot be excluded, serious adverse events including overdose have not been documented.

   5.4. Drug Accountability Study specific prescriptions can be used for dispensing the study product. The study medication can only be prescribed by qualified physicians clearly given this role on the study delegation log. Only people designated by the Principal Investigator (PI) can collect medication. Only PEA supplied for this study can be dispensed against the study specific prescription. Full accountability records will be completed including recording the batch, expiry date, people dispensing/checking the prescription, quantity and date of drug returns, empty packaging. Nothing is destroyed without the authorization from the PI.

   5.5. Storage of study medication PEA will be stored at room temperature (< 25 °C) and not kept in a refrigerator, in compliance with local regulations. It will be stored in a secure area away from other treatments and clearly marked for this study.

   Removal of study medication outside of expiry date/at trial conclusion and destruction 5.6. The expiry date will always be reported on the study medication. Study medication outside of the expiry date will not be dispensed and will be destroyed, subject to authorization, on an ongoing basis.

   5.7. Withdrawal of Subjects According to Declaration of Helsinki, all participants will have the right to withdraw from the study at any time without giving any reason, without any prejudice to their future medical care, and will be informed as such before consent. A participant's withdrawal will be discussed in terms of only discontinuing the study treatment and continuing follow-up visits. Should the patient request to completely withdraw from the study, the decision will be respected. All reasonable efforts will be made to ascertain the reason for discontinuation, even though participants will be not obliged to give any explanations. Already collected data will be kept and included in the final analysis. The investigator themselves may also withdraw participants for various reasons, including but not limited to the following: protocol violations, inter-current illness, adverse events, serious adverse events, suspected unexpected serious adverse reactions, administrative reasons, participation in the trial affecting their ongoing care, symptomatic worsening. In the latter case, participants will be followed up with the same schedule of research assessments as those who continue in the study, till they complete the 12-week follow-up period or till they progress to frank psychiatric disturbance (whichever is earlier). In case of autistic individuals experiencing progression to a full-blown psychiatric disorder, they will exit from the study intervention, be deemed as treatment failure, and will only be assessed for safety outcomes until they complete the 12-week follow-up period.

   5.8. Subject Compliance Pill-counts will be performed at FUP visits 1, 2, 3, and 4, in order to assess compliance with PEA treatment. Participants will be defined as complying in the presence of a pill count greater than 50% the expected number taken. Participants who are defined as non-complying with the medication will be coded as protocol deviators.

   5.9. Concomitant Medication Based on participants' clinical history, concomitant requirement of psychotropic medication is an exclusion criterion for the study, with the exception of patients undergoing Selective Serotonin Reuptake Inhibitor (SSRI) stable monotherapy (at least 8 months). Patients requiring continued treatment with other classes of psychotropic medications during the treatment phase may be withdrawn from the study by the PI. Very short-term treatment with rescue medications that have a well-established sedative or calming effect (e.g., Benzodiazepines) during the study may be allowed. Throughout the study, any other concomitant medications or treatments deemed necessary to provide adequate supportive care may be prescribed by investigators. A record will be kept to list all concomitant medications received during the treatment phase.
6. VISIT ASSESSMENTS

   The following visit assessments will be performed:

   6.1. First Screening Visit This will take place approximately one week prior to the Second Screening Visit and two to three weeks prior to the Baseline Visit. First, informed consent will be obtained from those who wish to take part to the study. Consenting patients will then be screened against the study inclusion and exclusion criteria and collecting information on their medical history. Individuals satisfying the criteria will be recruited by employed or delegated investigators. Also, consent will be obtained on all participants screened to collect plasma/serum/urine/fecal samples for routine biochemistry and haematology, endocannabinoid, immune, metabolic, and gut microbiome analysis. Consent will be sought to analyse screening data as well as regarding long-term follow-up beyond the outcomes of the trial and to link participants' data to routinely collected data sources such as Hospital Episode Statistics and General Practitioner records.

   6.2. Second Screening Visit This will take place one to two weeks prior to Baseline Visit. Safety blood and urine samples (for routine biochemistry and haematology) will be obtained, physical examination and vital signs will be recorded.

   6.3. Baseline Visit (day 0) Following satisfactory completion of screening, baseline measures (SCL-90-R, HADS, WHODAS-2.0), physical examination, blood, and fecal samples for endocannabinome (eCBome), immune, metabolic, and gut microbiota analyses will be acquired. Participants will be prescribed PEA and the medication will be dispensed. Side effects will also be assessed, by using the UKU side-effect rating scale.

   6.4. FUP Visit 1 (Week 4 ± 7 days, approximately day 28) This visit will be carried out at Month 1 and involve blood and fecal sampling for eCBome, immune, metabolic, and gut microbiota analyses, monitoring of compliance, side effects [39], adverse events, and dispensing of study medication.

   6.5. FUP Visit 2 (Week 12 ± 14 days, approximately Day 84) This visit will be carried out at Month 3 and involve clinical measures (SCL-90-R, HADS, WHODAS-2.0), physical examination, safety blood and urine samples, blood and fecal sampling for eCBome, immune, metabolic, and gut microbiota analyses, monitoring of compliance, side effects, adverse events, and dispensing of study medication.

   6.6. FUP Visit 3 (Week 24 ± 14 days, approximately Day 168) This visit will be carried out at Month 6 on those enrolled in the extension phase and involve, blood and fecal sampling for eCBome, immune, metabolic, and gut microbiota analyses, monitoring of compliance, side effects [39], adverse events, and dispensing of study medication.

   6.7. FUP Visit 4 (Week 36 ± 14 days, at approximately Day 252) This visit will be carried out at Month 9 on those enrolled in the extension phase and involve clinical measures (SCL-90-R, HADS, WHODAS-2.0), physical examination, safety blood and urine samples, blood and fecal sampling for eCBome, immune, metabolic, and gut microbiota analyses, monitoring of compliance, side effects, adverse events, and dispensing of study medication.

   6.8. Laboratory Tests Clinical Laboratory measures: blood tests for haematology (Full blood count and Haemoglobin), biochemistry (Urea & Electrolytes, liver function test, lipid profile), and immune profile characterization will be carried out at the clinical research recruitment hub as per their standard procedure. Blood results will be printed and filed as source in the patient folder. Serum samples for performing metabolic fingerprinting by Raman Spectroscopy, as well as blood and fecal samples for measurement of the levels of eCBome mediators and determination of the microbial composition in feces by Next Generation Sequencing (NGS) of 16SRNA and shotgun metagenomics methodologies, will be shipped to counseling specialized centers (e.g., Institute of Biomolecular Chemistry, Department of Chemical Sciences and Materials Technologies, National Research Council (CNR) Pozzuoli, Italy) where they will be stored and analysed.
7. SAMPLE SIZE 7.1. Proposed sample size We aim at enrolling 20 volunteers within 12 months from the start of recruitment.

   Sample size justification The number is coherent with suggested sample sizes for pilot studies and is deemed sufficient to evaluate feasibility outcomes. No powered sample size calculation was implemented for the pilot study.
8. METHODS 8.1. Data collection, management and archiving Assessment and collection of baseline, outcome and other trial data will be performed according to Visit assessments flow-chart. In case of trial intervention discontinuation, follow-up data will be collected anyway, unless a participant expresses the wish to be completely withdrawn from the study. All data source will be held on as a paper source data worksheet (SDW). These will be managed locally under the care of the recruiting and consenting site PI. Collected data will be held on paper SDW which will be thereafter recorded by allowed study team members on a 24-hour-accessible electronic-based data entry system hosted by the clinical research recruitment hub at ASUFC and University of Udine, consenting data entry to run in parallel with participant enrolment and visits. At the conclusion of the trial the study team will have resolved the data queries and request to remove user access to ensure that the final dataset cannot be changed. SDWs, electronic-based data, and the final statistical report will be archived. Systems will be in place to secure the data collection system against permanent loss and allow the recovery and restoration in the event of such a loss occurring.

   8.2. Data verification, statistical monitoring and analysis At the study start, a structured data verification plan will be agreed and developed by the Head Statistician of the research team. Data will be checked for consistency across paper- and electronic-based entry systems. Statistical monitoring will include the subject's severity level, eventual withdrawals, baseline data, FUP visits data, and AEs. The research team will approve a Statistical Analysis Plan within the early stages of the study, and before the Head Statistician summarizes any data. Proportions will be presented for each feasibility outcome. Interim analyses are not planned. The Head Statistician will both carry out and interpret statistical analysis. Our primary analysis will involve a generalized linear model with SCL-90-R symptom severity as the dependent measure and time as a repeated measure within subject. We are interested in whether there is a significant benefit over time with PEA treatment. WHODAS-2.0 and HADS ratings will be analysed in a similar manner. We will also conduct paired t tests based on baseline and endpoint assessments to examine measures of SCL-90-R severity and secondary measures. Rates of side effects will be reported, as well as reasons for dropouts from the trial.

   8.3. Missing Data We expect withdrawn participants to be missing at random, and very few participants withdrawing consent. All participants having at least one post-baseline outcome measure, would be included in each analysis. Nonetheless, patterns of missing data will be explored to investigate any evidence against missing at random, whose impact on the analysis will be considered by introducing imputation methods.
9. ETHICS 9.1. Ethics & Regulatory Approvals The trial will be conducted in accordance with the principles of the Declaration of Helsinki (1996) [48, 49], the principles of Good Clinical Practice (GCP) [50], and with all applicable regulatory requirements. This protocol and related documents will be submitted for review to the local Research Ethics Committee (REC).

   9.2. Consent Prior to Screening Those expressing interest into the study will be referred to the clinical research recruitment hub by their consultants. At screening, investigators will introduce the trial and provide the patients with exhaustive Patient Information Sheets (PIS). Allowed qualified physicians will discuss the trial with patients in light of the information provided in the PIS and give appropriate time for the participants to understand the information provided, before asking written informed consent from those willing to take part to the trial.

   9.3. Biological Samples The collection of routine blood samples, urine samples, fecal samples, and genotyping will be specifically addressed through the collection of ad hoc consent for biological materials. After collection at the research recruitment hub, obtained blood samples for haematology, biochemistry, and Immune profile characterization will be delivered by the study research team to the local laboratory for analysis. Blood and fecal samples collected to perform metabolic fingerprinting, measurement of the levels of eCBome mediators, and determination of the microbial composition, will be stored in local facilities under adequate conditions (-80°C) and then shipped to counseling specialized centers (e.g., Institute of Biomolecular Chemistry, Department of Chemical Sciences and Materials Technologies, National Research Council (CNR) Pozzuoli, Italy) for subsequent analysis.
10. CONFIDENTIALITY All study-related information will be stored securely at the study site. All participant information will be stored in locked file cabinets in areas with limited access. All laboratory specimens, reports, data collection, process, and administrative forms will be identified by a coded identification (ID) number only to maintain participant confidentiality. All records that contain names or other personal identifiers, such as locator forms and informed consent forms, will be stored separately from study records identified by code number. All local databases will be secured with password-protected access systems. Forms, lists, logbooks, appointment books, and any other listings that link participant ID numbers to other identifying information will be stored in a separate, locked file in an area with limited access. Participants' study information will not be released outside of the study without the written permission of the participant.
11. INSURANCE POLICY INFORMATION We did not deem it necessary to arrange a specific insurance policy for the present study. Any allergic reactions to PEA or unexpected adverse effects will be monitored when PEA is first administered at the Day Hospital service, which provides insurance coverage for patients admitted and undergoing non-invasive procedures as part of clinical routine.
12. DISSEMINATION POLICY The results of the study are intended to be reported and disseminated at national/international conferences and in peer-reviewed scientific journals. Our objective is to submit for publication the main results of the trial within two years of last patient recruitment.

ELIGIBILITY:
Inclusion Criteria:

* Individuals diagnosed with Level 1 ASD, as defined using Diagnostic and Statistical Manual of Mental Disorders-Fifth Edition (DSM-5);
* Aged 18-35 years;
* To be able to understand and communicate in Italian;
* To be able to give informed consent.

Exclusion Criteria:

* Level 2 or Level 3 ASD, as defined using Diagnostic and Statistical Manual of Mental Disorders-Fifth Edition (DSM-5) [47];
* Current diagnosis of a co-occurring major psychiatric disorder (e.g., major depressive disorder, bipolar affective disorder, psychotic disorders);
* Active suicidal ideation indicating significant current risk or history of serious suicide attempt in the opinion of the PI, as evaluated at the screening stage;
* Lifetime neurological disorders (e.g., epilepsy, except febrile convulsions) or severe intercurrent physical illness;
* Current treatment with psychotropic medication, with the exception of Selective Serotonin Reuptake Inhibitor (SSRI) stable monotherapy (at least 8 months);
* IQ < 70;
* Female patients who are pregnant, lactating or not using an acceptable effective form contraception if they are at risk of falling pregnant;
* Taking part in another pharmacological trial.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Symptom-Checklist-90-R | 12 weeks for the initial phase, further 24 weeks for the extension phase
  Global improvement in symptom intensity and psychological distress associated with autism through the Global Score Index (GSI) of the SCL-90-R

SECONDARY OUTCOMES:
World Health Organization Disability Assessment Schedule 2.0 | 12 weeks for the initial phase, further 24 weeks for the extension phase
  Impact on levels of personal autonomy as measured through the WHODAS 2.0 total score
Hospital Anxiety and Depression Scale | 12 weeks for the initial phase, further 24 weeks for the extension phase
  Severity of anxiety symptoms as assessed using the HADS
Symptom-Checklist-90-R | 12 weeks for the initial phase, further 24 weeks for the extension phase
  Severity of the somatisation, anxiety and depression subscales of the SCL-90-R
World Health Organization Disability Assessment Schedule 2.0 | 12 weeks for the initial phase, further 24 weeks for the extension phase
  Severity of neurocognitive and interpersonal functioning as assessed using the subdomains 1 'cognitive activities' and 4 'interpersonal relationships' of the WHODAS 2.0

CONTACTS AND LOCATIONS:
Overall Officials: Marco Colizzi, MD, PhD, Principal Investigator — Unit of Psychiatry, Department of Medicine (DAME), University of Udine (UNIUD)
Locations (1):
- Unit of Psychiatry, University Hospital of Udine, Udine, UD, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bortoletto R, Piscitelli F, Candolo A, Bhattacharyya S, Balestrieri M, Colizzi M. Questioning the role of palmitoylethanolamide in psychosis: a systematic review of clinical and preclinical evidence. Front Psychiatry. 2023 Jul 18;14:1231710. doi: 10.3389/fpsyt.2023.1231710. eCollection 2023. PMID 37533892
- [Result] Colizzi M, Bortoletto R, Costa R, Zoccante L. Palmitoylethanolamide and Its Biobehavioral Correlates in Autism Spectrum Disorder: A Systematic Review of Human and Animal Evidence. Nutrients. 2021 Apr 18;13(4):1346. doi: 10.3390/nu13041346. PMID 33919499
- [Result] Colizzi M, Bortoletto R, Colli C, Bonomo E, Pagliaro D, Maso E, Di Gennaro G, Balestrieri M. Therapeutic effect of palmitoylethanolamide in cognitive decline: A systematic review and preliminary meta-analysis of preclinical and clinical evidence. Front Psychiatry. 2022 Oct 28;13:1038122. doi: 10.3389/fpsyt.2022.1038122. eCollection 2022. PMID 36387000
- [Result] Bortoletto R, Balestrieri M, Bhattacharyya S, Colizzi M. Is It Time to Test the Antiseizure Potential of Palmitoylethanolamide in Human Studies? A Systematic Review of Preclinical Evidence. Brain Sci. 2022 Jan 12;12(1):101. doi: 10.3390/brainsci12010101. PMID 35053844
- [Result] Khalaj M, Saghazadeh A, Shirazi E, Shalbafan MR, Alavi K, Shooshtari MH, Laksari FY, Hosseini M, Mohammadi MR, Akhondzadeh S. Palmitoylethanolamide as adjunctive therapy for autism: Efficacy and safety results from a randomized controlled trial. J Psychiatr Res. 2018 Aug;103:104-111. doi: 10.1016/j.jpsychires.2018.04.022. Epub 2018 May 1. PMID 29807317